CLINICAL TRIAL: NCT02139358
Title: Phase I/IIa Trial of Gemcitabine Plus Trastuzumab and Pertuzumab in Previously Treated Metastatic HER2+ Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17656; ML28939 (Other: Genentech)
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: Breast - Female; Metastatic; HER2+
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation / Phase II Treatment (Experimental): Single arm, non-randomized, open label phase I/II multisite Simon two stage minimax trial. Gemcitabine plus trastuzumab and pertuzumab.
  Interventions: Drug: Gemcitabine; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Gemcitabine — The Phase I trial will start at the recommended phase II dose (RP2D) for gemcitabine but will have a de-escalation dose levels in the event that an unacceptable toxicity requires dose reduction. Dose level 0 = gemcitabine (1200 mg/m2) IV D1,8 q21 days; Dose level -1 = gemcitabine (1000 mg/m^2) IV D1,8 q21 days; Dose level -2 = gemcitabine (850 mg/m^2) IV D1,8 q21 days. The RP2D will be the dose level where 0-1 dose limiting toxicities (DLTs) in six patients occur.
  Other Names: GEMZAR®
Drug: Trastuzumab — Trastuzumab will be given using an 8 mg/kg loading dose on cycle one, day one (C1D1), followed by 6 mg/kg IV on subsequent cycles every (q) 21 days.
  Other Names: Herceptin®
Drug: Pertuzumab — Pertuzumab will be given using an 840 mg IV loading dose on C1D1, followed by 420 mg IV on subsequent cycles q 21 days.
  Other Names: PERJETA®

SUMMARY:
The purpose of this study is to evaluate the safety and activity of gemcitabine plus trastuzumab and pertuzumab in patients with metastatic human epidermal growth factor receptor 2 (HER2)+ breast cancer who have progressed on at least one prior line of chemotherapy plus HER2 targeted agent such as T-DM1, trastuzumab, or lapatinib.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females (aged 18 or older) with histologically confirmed, metastatic human epidermal growth factor receptor 2 (HER2)+ (by immunohistochemistry (IHC) 3+ or fluorescence in situ hydridization (FISH) ratio ≥ 2.0) breast cancer
* Have progressed on at least one prior line of chemotherapy plus HER2 directed therapy such as trastuzumab and/or pertuzumab in the metastatic setting. T-DM1 would count as a line of therapy and patients previously treated with T-DM1 are eligible.
* Have not been treated with gemcitabine in the metastatic setting
* Measurable disease per Response Evaluation in Solid Tumors (RECIST) 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 2≤
* Left Ventricular Ejection Fraction (LVEF) ≥ 50% at baseline as determined by either echocardiogram (ECHO) or multiple gated acquisition scan (MUGA)
* Adequate bone marrow function as indicated by the following: absolute neutrophil count (ANC) >1500/µL; Platelets ≥100,000/µL; Hemoglobin >10 g/dL
* Adequate renal function, as indicated by creatinine ≤1.5x upper limit of normal (ULN)
* Adequate liver function, as indicated by bilirubin ≤1.5x ULN, aspartic transaminase (AST) or alanine transaminase (ALT) <2x ULN unless related to metastatic breast cancer to the liver (in which case AST/ALT < 5x ULN is allowed).
* Signed informed consent
* Adequate birth control in sexually active women of childbearing potential

Exclusion Criteria:

* Active uncontrolled infection or major concurrent illness which in the opinion of the investigator would render the participant unsafe to proceed with the study
* Uncontrolled central nervous system (CNS) metastases. Treated, non-progressing CNS disease (documented by brain magnetic resonance imaging [MRI]) off corticosteroids for at least 1 month potential participants are eligible.
* Women who are pregnant or lactating
* Prior chemotherapy within the last 3 weeks (last 6 weeks for nitrosureas/mitomycin)
* Prior radiation therapy within the last 4 weeks; prior radiation therapy to indicator lesion (unless objective disease recurrence or progression within the radiation portal has been documented since completion of radiation)
* Other concomitant active malignancies
* History of significant cardiac disease, cardiac risk factors or uncontrolled arrhythmias
* Ejection fraction <50% or below the lower limit of the institutional normal range, whichever is lower
* Hypersensitivity to any of the study medications
* Untreated psychiatric conditions preventing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Soliman, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center October 2014 through October 2016.
Groups:
- Dose Escalation / Phase II Treatment: Single arm, non-randomized, open label phase I/II multisite Simon two stage minimax trial. Gemcitabine plus trastuzumab and pertuzumab.
  Gemcitabine: The Phase I trial will start at the recommended phase II dose (RP2D) for gemcitabine but will have a de-escalation dose levels in the event that an unacceptable toxicity requires dose reduction. Dose level 0 = gemcitabine (1200mg/m2) IV D1,8 q21 days; Dose level -1 = gemcitabine (1000 mg/m^2) IV D1,8 q21 days; Dose level -2 = gemcitabine (850 mg/m^2) IV D1,8 q21 days. The RP2D will be the dose level where 0-1 dose limiting toxicities (DLTs) in six patients occur.
  Trastuzumab: Trastuzumab will be given using an 8 mg/kg loading dose on cycle one, day one (C1D1), followed by 6 mg/kg IV on subsequent cycles every (q) 21 days.
  Pertuzumab: Pertuzumab will be given using an 840 mg IV loading dose on C1D1, followed by 420 mg IV on subsequent cycles q21 days.
Period: Overall Study
Arm/Group | Dose Escalation / Phase II Treatment
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Dose Escalation / Phase II Treatment
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 58.2 [46 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Recommended Phase II Dose (RP2D)
Description: The RP2D dose in mg/m^2 of gemcitabine along with standard doses of pertuzumab (840 mg loading/420 mg maintenance) and Herceptin (8 mg/kg loading, 6 mg/kg maintenance). Safety data to be described using Common Terminology Criteria for Adverse Events (CTCAE) 4.0 terminology. Any participant who receives any dose of the study treatment will be evaluated for the safety/toxicity endpoints in the trial.
Time Frame: 6 Months
Population: All participants enrolled during Phase 1
Measure: Number; unit: dose in mg/m^2
Arm/Group | Dose Escalation / Phase II Treatment
Number analyzed (Participants) | 6
dose in mg/m^2 | 1200

2. Primary Outcome: Phase II: Objective Response Rate (ORR)
Description: Objective Response Rate: Response according to Response Evaluation in Solid Tumors (RECIST) 1.1 for the combination of gemcitabine+trastuzumab+pertuzumab at the recommended phase II dose. Complete Response (CR): Disappearance of all evidence of tumor for at least two cycles of therapy. Tumor markers must be normal. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter of target lesions, taking a reference the baseline sum longest diameter. Stable Disease (SD): Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started. Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the beginning of treatment or the appearance of one or more new lesions.
Time Frame: Up to 36 Months
Population: All participants who have undergone 2 treatment cycles followed by a response scan and have documented best response data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation / Phase II Treatment
Number analyzed (Participants) | 10
Participants
  Complete Response | 1
  Partial Response | 1
  Stable Disease | 8

3. Secondary Outcome: Phase II: Progression Free Survival (PFS)
Description: Median progression free survival (in months) for all participants evaluable for response. The time-to-event data will be summarized using Kaplan-Meir curve method for all patients who are evaluable for the ORR endpoint. Progressive disease (PD): At least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the beginning of treatment or the appearance of one or more new lesions.
Time Frame: Up to 12 months
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation / Phase II Treatment
Number analyzed (Participants) | 15
months | 6.4883 [2.7807 to 9.0372]

4. Secondary Outcome: Overall Survival (OS)
Description: Median overall survival (in months) for all participants evaluable for response. The length of time from the start of treatment that participants are still alive.
Time Frame: Up to 36 months
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation / Phase II Treatment
Number analyzed (Participants) | 15
months | 11.3545 [6.2897 to 14.0028]

ADVERSE EVENTS:
Time Frame: 3 years, 7 months
Arm/Group | Dose Escalation / Phase II Treatment
All-Cause Mortality (participants affected / at risk) | 2/15
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation / Phase II Treatment (N=15)
Cardiac arrest (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Sudden death NOS (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation / Phase II Treatment (N=15)
Neutrophil count decreased (Investigations) | 12 (47)
Lymphocyte count decreased (Investigations) | 10 (19)
Platelet count decreased (Investigations) | 9 (24)
White blood cell decreased (Investigations) | 9 (48)
Alanine aminotransferase increased (Investigations) | 6 (12)
Aspartate aminotransferase increased (Investigations) | 6 (17)
Alkaline phosphatase increased (Investigations) | 2 (3)
Creatinine increased (Investigations) | 1 (2)
Ejection fraction decreased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (13)
Nausea (Gastrointestinal disorders) | 9 (11)
Vomiting (Gastrointestinal disorders) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 10 (12)
Infusion related reaction (General disorders) | 3 (3)
Pain (General disorders) | 3 (4)
Edema limbs (General disorders) | 2 (3)
Fever (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (8)
Hypokalemia (Metabolism and nutrition disorders) | 5 (10)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 11 (39)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Right wrist swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Left chest wall - Abnormal sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Papulopustular rash (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (5)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Cervical polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified and polyps) - Other, Goiter with thyroid modules (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT02139358/Prot_SAP_000.pdf